CLINICAL TRIAL: NCT04175145
Title: Impact of Metal Density on Deformity Correction in Posterior Fusions for Adolescent Idiopathic Scoliosis
Brief Title: Impact of Metal Density on Deformity Correction for Adolescent Idiopathic Scoliosis
Status: Completed | Type: Observational
Sponsor: Ghurki Trust and Teaching Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 19
Record Dates: First submitted 2019-11-11; First posted 2019-11-22 (Actual); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Adolescent Idiopathic Scoliosis
Keywords: Adolescent idiopathic scoliosis; posterior instrumentation; metal density; correction; Pakistan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Posterior spinal instrumentation — A fusion construct consisting of all pedicle screws except at uppermost instrumented vertebra. Contoured dual 6-mm stainless steel rods were used to connect the construct. Pedicle screw location and density was determined by the surgeon based on perceived curve stiffness and fusion length with an even distribution of fixation points along the construct. Pedicle screw instrumentation was performed by the free hand technique with biplanar fluoroscopic and direct screw EMG impedance testing for confirmation of placement. Reduction was via cantilever-segmental-translation maneuver in all cases.

SUMMARY:
A retrospective analysis to ascertain the correlation between metal density and deformity correction among individuals with adolescent idiopathic scoliosis.

DETAILED DESCRIPTION:
Posterior spinal fusion with pedicle screws has become the "gold standard" for the management of adolescent idiopathic scoliosis (AIS). Pedicle screws provide three column fixation through the strongest part of vertebra thereby enhancing surgeon's ability to do a 3-dimensional deformity correction. The higher pullout strength results in less long-term loss of correction, shorter fusions resulting in preservation of motion segments, lower pseudarthrosis rates and lower implant failures compared with these alternative posterior instrumentation systems. However, studies are contradictoryregarding the effect of metal density on coronaland sagittal curve corrections. Multiple factors including curve flexibility, instrumentation and rod types, reduction strategies and curve types, affect outcomes. Given this, intraoperative decisions regarding the number of anchorage points remain difficult, with considerable inter-surgeon variability.

The rationale for using a high implant density constructs is to obtain more rigid fixation and to limit potential stress concentration at any one screw. Furthermore, health-related quality of life instruments such as the SRS 22, 24, or 30 seem to show little correlation with curve correction. The placement of every additional pedicle screw is associated with increased operative time, risk of neurological deterioration and increased implant cost. If implant density can be lowered without compromising clinical results, reducing the number of screws may improve the efficiency and cost effectiveness of scoliosis surgery. Several authors have demonstrated successful results with low-density instrumentation for the treatment of scoliosis. The purpose of this retrospective review is to describe the demographics of our patient population and to ascertain correlation between metal density and correction achieved.

ELIGIBILITY:
Inclusion Criteria:

* Patients with adolescent idiopathic scoliosis
* Age more than 10 years at time of surgery
* Posterior instrumentation consisting of all pedicle screw construct except for bilateral hooks at the uppermost instrumented vertebra
* A major curve magnitude between 45 and 80 degrees.

Exclusion Criteria:

* Scoliosis patients with a diagnosis other than adolescent idiopathic scoliosis
* Previous spine surgery
* Use of spinal osteotomies in addition to posterior spinal fusion with pedicle screws
* ALenke 5 curve
* Patients with less than 2 years' follow-up
* Use of hooks or wires below the uppermost instrumented level

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Retrospective review of all patients with Adolescent Idiopathic Scoliosis patients operated at our hospital during study period
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Degree of correction achieved | 2 years
  (Preop Cobb angle - Postop Cobb angle/ Preop Cobb angle * 100)
Cobb angle | 2 years
  Cobb angle is measured as angle sub-tented between the upper and lower end vertebrae (end vertebrae is defined as the vertebra that is most tilted from the horizontal apical vertebra)

CONTACTS AND LOCATIONS:
Overall Officials: Dr Irfan Qadir, Principal Investigator — Department of Orthopaedics and Spine Surgery, Ghurki Trust Teaching Hospital; Prof.Amer Aziz, Professor and Chief, Study Director — Department of Orthopaedics and Spine Surgery, Ghurki Trust Teaching Hospital; Abdullah Shah, Assistant Professor, Study Chair — Department of Orthopaedics and Spine Surgery, Ghurki Trust Teaching Hospital; Syed Roman Alam, Resident, Study Chair — Department of Orthopaedics and Spine Surgery, Ghurki Trust Teaching Hospital; Haseeb Hussain, Senior Registrar, Study Chair — Department of Orthopaedics and Spine Surgery, Ghurki Trust Teaching Hospital; Prof.Rizwan Akram, Professor, Study Chair — Department of Orthopaedics and Spine Surgery, Ghurki Trust Teaching Hospital

IPD SHARING:
Plan to Share IPD: No